CLINICAL TRIAL: NCT00428064
Title: A Randomized, Open-Label Study of Continuous Therapy With Cyclosporine and Sirolimus Versus Induction With Cyclosporine and Sirolimus Followed by Continuous Therapy With Sirolimus in Renal Allograft Recipients
Brief Title: Study Evaluating Sirolimus and Cyclosporine in Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0468H1-310
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2007-01

CONDITIONS: Renal Transplantation
Keywords: Renal allograft; Renal; Kidney; Transplant
MeSH Terms: interventions — Sirolimus; Cyclosporine

INTERVENTIONS:
Drug: Sirolimus
Drug: cyclosporine

SUMMARY:
To assess equivalence in the rates of functional graft survival at 12 months after transplantation in patients receiving continuous therapy with cyclosporine (CsA, Sandimmune, Neoral) and sirolimus versus induction with CsA and sirolimus followed by CsA elimination and concentration-controlled sirolimus.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease, with patients receiving a primary or secondary renal allograft from a cadaveric donor, from a living-unrelated donor, or from a living-related (excluding 0 antigen mismatch) donor.
* Women who are of childbearing potential must have a negative pregnancy test before sirolimus administration and agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months following discontinuation of sirolimus

Exclusion Criteria:

* Evidence of active systemic or localized major infection at the time of initial sirolimus administration
* Evidence of infiltrate, cavitation, or consolidation on chest x-ray obtained during pre-study screening.
* Chronic antiarrhythmic therapy for ventricular arrhythmia or other cardiac abnormality contraindicating general anesthesia or surgery

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408
Dates: Start 1998-05; Study Completion 2004-06

PRIMARY OUTCOMES:
Equivalence of graft survival at month 12

SECONDARY OUTCOMES:
Renal function; biopsy-confirmed acute rejection, grade of acute rejection; subject and graft survival; incidence of infection, malignancy, treatment failure, and of chronic rejection as determined by protocol biopsies; quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Friend P, Russ G, Oberbauer R, Murgia MG, Tufveson G, Chapman J, Blancho G, Mota A, Grandaliano G, Campistol JM, Brault Y, Burke JT; Rapamune Maintenance Regimen (RMR) Study Group. Incidence of anemia in sirolimus-treated renal transplant recipients: the importance of preserving renal function. Transpl Int. 2007 Sep;20(9):754-60. doi: 10.1111/j.1432-2277.2007.00506.x. Epub 2007 Jun 12. PMID 17565578